CLINICAL TRIAL: NCT05486936
Title: RapidPlan Models Establishment for Node-Positive Breast Cancer Treated With Hypofractionation Using Edge/Truebeam
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, JIAYI CHEN, Chief of Department of Radiation Oncology, Ruijin Hospital
Other Study IDs: RJrapidplan
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
Keywords: hypofractionated radiotherapy; IMRT; internal mammary nodes; rapidplan model
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study arm: Eligible breast cancer patients will receive hypofractionated radiotherapy of 2.67 Gy for 16 fractions (and sequential tumor bed boost of 2.67 Gy for 4 fractions in patients with intact breast) to ipsilateral chest wall or whole breast and regional lymph regions (including supraclavicular and internal mammary lymph nodes) at the discrection of radition oncologists. The plans which pass the on-line verification will then be de-identified and transferred to RapidPlan configuration workspace for RNI model training and verification.All enrolled patients will be regularly followed up during and after RT. Acute and late toxicity will be documented as well as tumor control endpoints.
  Interventions: Radiation: hypofractionated radiation

INTERVENTIONS:
Radiation: hypofractionated radiation — Eligible breast cancer patients will receive hypofractionated radiotherapy of 2.67 Gy for 16 fractions (and sequential tumor bed boost of 2.67 Gy for 4 fractions in patients with intact breast) to ipsilateral chest wall or whole breast and regional lymph regions (including supraclavicular and internal mammary lymph nodes) at the discrection of radition oncologists.

SUMMARY:
The purpose of this trial is to establish a feasible DVH estimation model of integrated IMRT plan for HF-RNI with Eclipse™ Treatment Planning System and a Varian RapidPlan™ model based on the above DVH constraints.

DETAILED DESCRIPTION:
Eligible breast cancer patients will receive hypofractionated radiotherapy of 2.67 Gy for 16 fractions (and sequential tumor bed boost of 2.67 Gy for 4 fractions in patients with intact breast) to ipsilateral chest wall or whole breast and regional lymph regions (including supraclavicular and internal mammary lymph nodes) at the discrection of radition oncologists. CTV including breast/chest wall and regional nodes will be contoured according to RTOG contouring atlas. Integrated multi-beam IMRT plan will be generated and optimized using our predefined protocol for OAR constrains and target coverage. All integrated IMRT plans will be designed using the Eclipse™ Treatment Planning System. All these tight margin IMRT plan will be passed in pre-treatment dry run with the motion management workflow involved and the target coverage during the treatment will be confirmed. The plans which pass the above on-line verification will then be de-identified and transferred to RapidPlan configuration workspace for RNI model training and verification.All enrolled patients will be regularly followed up during and after RT. Acute and late toxicity will be documented as well as tumor control endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years old
* Ipsilateral clinically diagnosed and histologically confirmed invasive breast cancer pT1-3
* ≥1 pathologically positive axillary lymph nodes
* Karnofsky Performance Status scoring ≥80
* Surgery wound healed without infection
* Anticipative overall survival >5 years
* Pathologically surgical margin >2mm
* ER (estrogen-receptor), PR (progesterone-receptor), HER2 (human epidermal growth factor receptor 2) and Ki67 testing can be performed on the primary breast tumor
* Women of child-bearing potential must agree to use adequate contraception for up to 1 month before study treatment and the duration of study participation
* Ability to understand and willingness to participate the research and sign the consent form

Exclusion Criteria:

* Axillary dissection of less than 10 lymph nodes
* Pathologically positive ipsilateral supraclavicular lymph node
* Pathologically or radiologically confirmed positive ipsilateral internal mammary lymph nodes
* Pregnant or lactating women
* Treated with breast reconstruction surgery
* Severe non-neoplastic medical comorbidities
* History of non-breast malignancy within 5 years with the exception of lobular carcinoma in situ, basal cell carcinoma of the skin, carcinoma in situ of skin and carcinoma in situ of the cervix
* simultaneous contralateral breast cancer
* Previous RT to the neck, chest and/or ipsilateral axillary region
* Active collagen vascular disease
* Definitive pathological or radiologic evidence of distant metastatic disease
* Primary T4 tumor
* Interval between radical surgery (mastectomy or breast conserving surgery) and radiotherapy was more than 12 weeks or interval between last dose of adjuvant chemotherapy and radiotherapy was more than 8 weeks

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited by radiation oncologists in outpatient department. For each potential participant, the background of this trial will be introduced by the clinicians or research nurses at their first visit.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
≥Grade 2 acute radiation-induced toxicity | 6 months
  Within time from beginning of radiotherapy to 6 months after completion of radiotherapy, any acute radiation-induced toxicity will be assessed every week during radiotherapy, 4 weeks, 3 months and 6 months after the last fraction received using the (Common Terminology Criteria for Adverse Events) CTCAE 3.0 and recorded.

SECONDARY OUTCOMES:
≥Grade 2 Late Radiation-induced Toxicity | 5 years
  Within time from 6 months after completion of radiotherapy to 5 years after completion of radiotherapy, any late toxicity will be assessed every 6 months during the first 2 years and annually thereafter using the RTOG/ (European Organization for Research on Treatment of Cancer) EORTC Late Radiation Morbidity Scoring Schema and CTCAE 3.0
Number of Participants with excellent or good Cosmetic outcomes following breast conserving surgery-Harvard/NSABP/RTOG scoring scale | 5 years
  The time from the date of randomization to 5 years after completion of radiotherapy, the cosmetic outcomes will be evaluated before radiotherapy, every week during radiotherapy, 4 weeks after the last fraction received, every 6 months during the first 2 years and annually thereafter. The cosmetic outcomes are evaluated based on the Allegheny General Modification of the Harvard/(National Surgical Adjuvant Breast and Bowel Project) NSABP/ (Radiation Therapy Oncology Group) RTOG scoring scale which graded patients into the following four classifications: excellent, when compared to the untreated breast, there is a minimal or no difference in the size or shape of the treated breast; good, slight difference in the size or shape of the treated breast; fair, obvious difference in the size or shape of the treated breast; and poor, marked change in the size or shape of the treated breast.
Quality of Life-EORTC QLQ-C30 and QLQ-BR23 | 1 years
  The time from the date of randomization to 5 years after completion of radiotherapy, Quality of life will be assessed before radiotherapy, every week during radiotherapy, 4 weeks after the last fraction received, every 6 months during the first 2 years and annually thereafter using self-administered questionnaire EORTC QLQ-C30 and QLQ-BR23.
Quality of Life-EORTC QLQ-C30 and QLQ-BR23 | 5 years
  The time from the date of randomization to 5 years after completion of radiotherapy, Quality of life will be assessed before radiotherapy, every week during radiotherapy, 4 weeks after the last fraction received, every 6 months during the first 2 years and annually thereafter using self-administered questionnaire EORTC QLQ-C30 and QLQ-BR23.
Locoregional recurrence (LRR) | 5 years
  Any first recurrence confirmed by histology or cytology within the ipsilateral chest wall and/or regional nodes area (including supraclavicular, infraclavicular or internal mammary lymph nodes)
distant metastasis free survival (DMFS) | 5 years
  The time from the date of randomization to any recurrence of tumor at distant sites or death from any cause.
invasive recurrence free survival (IRFI) | 5 years
  The time from the date of randomization to any invasive recurrence of tumor or death from any cause.
overall survival (OS) | 5 years
  The time from the date of randomization to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Chen, MD, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China